CLINICAL TRIAL: NCT05128942
Title: A Phase 2 Study to Evaluate the Safety, Efficacy and Pharmacokinetics of SPR001 (Tildacerfont) in Children Aged 2 to 17 Years With Congenital Adrenal Hyperplasia (CAH)
Brief Title: A Phase 2 Study to Evaluate the Safety, Efficacy and PK of Tildacerfont in Children Aged 2-17 Years With CAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The SPR001-203 clinical trial did not achieve the primary efficacy endpoint of the absolute change in daily GC dose from baseline at week 24. It was decided to terminate the SPR001-205 in response to the SPR001-203 efficacy data.
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPR001-205
Record Dates: First submitted 2021-10-27; First posted 2021-11-22 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Congenital Adrenal Hyperplasia; 21-OHD
Keywords: Pediatric; CAH; Adrenal Disorder; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Adrenal Gland Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to treatment cohorts by age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: Age 11-17 Treatment with Tildacerfont (Experimental): 50 mg daily for 12 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 2: Age 11-17 Treatment with Tildacerfont (Experimental): 200 mg daily for 12 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 3: Age 2-10 Treatment with Tildacerfont (Experimental): 50, 100, or 200 mg daily for 12 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 4: Age >/= 18 Treatment with Tildacerfont (Experimental): 200 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 5: Age >/= 18 Treatment with Tildacerfont (Experimental): 300 or 400 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 6: Age 11-17 Treatment with Tildacerfont (Experimental): 200 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 7: Age 2-10 Treatment with Tildacerfont (Experimental): 200 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 8: Age 11-17 Treatment with Tildacerfont (Experimental): 300 or 400 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont
- Cohort 9: Age 2-10 Treatment with Tildacerfont (Experimental): 300 or 400 mg twice daily for 4 consecutive weeks.
  Interventions: Drug: Tildacerfont

INTERVENTIONS:
Drug: Tildacerfont — Oral tablet formulation taken once daily in combination with glucocorticoid therapy.
  Other Names: SPR001

SUMMARY:
An investigation of the safety and efficacy of tildacerfont in participants with CAH.

DETAILED DESCRIPTION:
This is a Phase 2 open-label study with up to 10 cohorts that will evaluate the safety, efficacy, and PK of different tildacerfont dosing regimens potentially up to 200mg QD for 12 weeks in children with classic CAH, and up to 400mg BID for 4 weeks in children and adults with classic CAH.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 2+
* Diagnosis of CAH due to 21-hydroxylase deficiency (OHD) and/or elevated 17- hydroxyprogesterone (OHP) requiring ongoing GC replacement since diagnosis
* Stable dose of GC replacement for at least 1 month prior to screening

Exclusion Criteria:

* History of bilateral adrenalectomy or hypopituitarism
* Clinically significant unstable medical conditions, illness, or chronic diseases
* History of active bleeding disorders

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Spruce Biosciences
Locations (13):
- United States (13):
  - Spruce Study Site, Sacramento, California
  - Spruce Study Site, San Diego, California
  - Spruce Study Site, Chicago, Illinois
  - Spruce Study Site, Minneapolis, Minnesota
  - Spruce Study Site, Buffalo, New York
  - Spruce Study Site, Providence, Rhode Island
  - Spruce Study Site, Columbia, South Carolina
  - Spruce Study Site, Dallas, Texas
  - Spruce Study Site, Edinburg, Texas
  - Spruce Study Site, Fort Worth, Texas
  - Spruce Study Site, Salt Lake City, Utah
  - Spruce Study Site, Charlottesville, Virginia
  - Spruce Study Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated before participants could be enrolled in Cohort 9
Pre-assignment Details: Doses in Cohort 3 were determined to be weight-based dose equivalents of >/= 200 mg QD. Upon completion of the 4-week dosing on participants from Cohorts 4&6, DMC assessed safety data and provided recommendations on dosing for Cohort 5 (initiated either at 300mg or 400mg BID) and for Cohort 7. Following completion of Cohorts 5&7, DMC reviewed safety data made recommendations on whether to proceed to Cohort 8 and at what dose for each participant (either 300mg or 400mg).
Groups:
- Cohort 4: Treatment With Tildacerfont; Cohort 6: Treatment With Tildacerfont; Cohort 7: Treatment With Tildacerfont: 200 mg twice daily for 4 consecutive weeks.
- Cohort 5: Treatment With Tildacerfont; Cohort 8: Treatment With Tildacerfont; Cohort 9: Treatment With Tildacerfont: 300 or 400 mg twice daily for 4 consecutive weeks.
Period: Overall Study
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont | Cohort 9: Treatment With Tildacerfont
Started | 7 | 7 | 18 | 2 | 6 | 8 | 12 | 7 | 0
Completed | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 17 | 2 | 5 | 8 | 12 | 7 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Termination by Sponsor | 2 | 6 | 14 | 2 | 4 | 8 | 11 | 6 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont | Total
Number analyzed (Participants) | 7 | 7 | 18 | 2 | 6 | 8 | 12 | 7 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.238 (1.688) | 14.381 (2.539) | 7.722 (2.3279) | 25.125 (8.8978) | 26.333 (8.2635) | 14.354 (2.0792) | 6.882 (2.5185) | 15.214 (1.7192) | 12.604 (6.7977)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 9 | 1 | 4 | 6 | 7 | 4 | 41
  Male | 0 | 4 | 9 | 1 | 2 | 2 | 5 | 3 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 7 | 1 | 3 | 2 | 3 | 2 | 21
  Not Hispanic or Latino | 6 | 5 | 11 | 1 | 3 | 6 | 9 | 5 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 7 | 5 | 14 | 0 | 6 | 7 | 12 | 7 | 58
  Other | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAE) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: To evaluate safety of tildacerfont in participants with CAH as measured by number of subjects with adverse events following dosing by CTCAE version 5.0
Time Frame: 12 weeks
Population: For Cohorts 5 and 8, the Statistical Analysis Plan pre-specified to analyze the data separately "per Cohort," without regard to dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont
Number analyzed (Participants) | 7 | 7 | 18 | 2 | 6 | 8 | 12 | 7
Participants | 4 | 6 | 18 | 2 | 3 | 8 | 12 | 5

2. Secondary Outcome: Proportion of Participants Who Achieve a Reduction in Androstenedione (A4) or Reduction in Glucocorticoid (GC) Dosing
Description: To determine the efficacy of tildacerfont on disease control or reduction of GC use in participants with classic CAH as measured by number of subjects who achieve a reduction in A4 or reduction in GC dosing during treatment period
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 7: Treatment With Tildacerfont; Cohort 8: Treatment With Tildacerfont: 300 or 400 mg twice daily for 4 consecutive weeks.
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont
Number analyzed (Participants) | 5 | 7 | 18 | 2 | 3 | 8 | 12 | 2
Participants | 5 | 4 | 14 | 2 | 0 | 4 | 1 | 0

3. Secondary Outcome: Proportion of Participants With Elevated Baseline A4 Who Achieve a Reduction in A4
Description: To determine the efficacy of tildacerfont on disease control in participants with classic CAH measured by the number of participants with elevated baseline A4 who achieve reduction in A4 at week 4
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont
Number analyzed (Participants) | 4 | 5 | 13 | 1 | 1 | 8 | 12 | 2
Participants | 4 | 3 | 9 | 0 | 1 | 6 | 5 | 0

4. Secondary Outcome: Proportion of Participants With Elevated Baseline A4 Who Achieve a Reduction in A4 Who Achieve A4 Normalization
Description: To determine the efficacy of tildacerfont on disease control in participants with classic CAH measured by the number of participants with elevated baseline A4 who achieve reduction in A4 at week 4 or week 12
Time Frame: 4 weeks or 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: Treatment With Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: Treatment With Tildacerfont
Number analyzed (Participants) | 4 | 5 | 13 | 1 | 1 | 8 | 12 | 2
Participants
  Week 4 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
  Week 12 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Cohort 5: 300 mg Tildacerfont; Cohort 8: 300 mg Tildacerfont: 300 mg twice daily for 4 consecutive weeks.
- Cohort 5: 400 mg Tildacerfont; Cohort 8: 400 mg Tildacerfont: 400 mg twice daily for 4 consecutive weeks.
Arm/Group | Cohort 1: Age 11-17 Treatment With Tildacerfont | Cohort 2: Age 11-17 Treatment With Tildacerfont | Cohort 3: Age 2-10 Treatment With Tildacerfont | Cohort 4: Treatment With Tildacerfont | Cohort 5: 300 mg Tildacerfont | Cohort 5: 400 mg Tildacerfont | Cohort 6: Treatment With Tildacerfont | Cohort 7: Treatment With Tildacerfont | Cohort 8: 300 mg Tildacerfont | Cohort 8: 400 mg Tildacerfont
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/18 | 0/2 | 0/1 | 0/5 | 0/8 | 0/12 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 1/18 | 0/2 | 0/1 | 0/5 | 0/8 | 1/12 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 4/7 | 6/7 | 18/18 | 2/2 | 0/1 | 3/5 | 8/8 | 12/12 | 2/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Age 11-17 Treatment With Tildacerfont (N=7) | Cohort 2: Age 11-17 Treatment With Tildacerfont (N=7) | Cohort 3: Age 2-10 Treatment With Tildacerfont (N=18) | Cohort 4: Treatment With Tildacerfont (N=2) | Cohort 5: 300 mg Tildacerfont (N=1) | Cohort 5: 400 mg Tildacerfont (N=5) | Cohort 6: Treatment With Tildacerfont (N=8) | Cohort 7: Treatment With Tildacerfont (N=12) | Cohort 8: 300 mg Tildacerfont (N=3) | Cohort 8: 400 mg Tildacerfont (N=4)
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | NA | 0 | 1 | 0 | NA
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Age 11-17 Treatment With Tildacerfont (N=7) | Cohort 2: Age 11-17 Treatment With Tildacerfont (N=7) | Cohort 3: Age 2-10 Treatment With Tildacerfont (N=18) | Cohort 4: Treatment With Tildacerfont (N=2) | Cohort 5: 300 mg Tildacerfont (N=1) | Cohort 5: 400 mg Tildacerfont (N=5) | Cohort 6: Treatment With Tildacerfont (N=8) | Cohort 7: Treatment With Tildacerfont (N=12) | Cohort 8: 300 mg Tildacerfont (N=3) | Cohort 8: 400 mg Tildacerfont (N=4)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7 | 0 | 0 | 1 | 1 | 5 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faece pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 9 | 1 | 0 | 0 | 1 | 4 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 5 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Beta hemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
17-hydroxyprogesterone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood androstenedione increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine output increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autism spectrum disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT05128942/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT05128942/SAP_003.pdf
  • Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT05128942/ICF_002.pdf